CLINICAL TRIAL: NCT00424658
Title: Sleep Apnea. Concordance Between Non-reference and Reference Centres
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: Sleep concordance; NCT00424879 (obsolete NCT alias)
Record Dates: First submitted 2007-01-17; First posted 2007-01-19 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2007-01

CONDITIONS: Sleep Apnea
Keywords: breathing disorders
MeSH Terms: conditions — Sleep Apnea Syndromes; Dyspnea

INTERVENTIONS:
Procedure: SAHS diagnosis

SUMMARY:
When a disorder is as prevalent as sleep apnea hypopnea syndrome various medical levels and strategies should be implicated. We to evaluate the degree of concordance in management between a sleep reference centre and non-reference centres.

DETAILED DESCRIPTION:
INTRODUCTION: When a disorder is as prevalent as SAHS, different medical levels should be involved to facilitate diagnosis for all patients, or at least those that are in moderate-severe or risk groups. A good option could be to transfer the patient assessment to non-reference centres (NRC). Therefore, the aim of the present study was to evaluate this strategy by analysing the degree of concordance between RC and NRC in treatment decision and management of SAHS patients.

MATERIALS AND METHODS: Study subjects: The study population consisted of 88 consecutive subjects with a suspicion of SAHS (age 50±11 years, 81 % male, BMI 30±4 K/m2) from the out-patient clinics of three NRC in the Barcelona area: Hospital Asil de Granollers, Hospital General de Vic and Hospital de Terrassa.

Study design: The patients were evaluated independently, at random, over the course of 1 month in the RC and NRC. In both types of centre, the patient evaluation was carried out on the basis of the clinical history, with a specific questionnaire about sleep disordered breathing, and a sleep study in the hospital. The evaluation was performed by a sleep physician in the RC and by a respiratory physician with training in sleep medicine in the NRC. In both cases, the choice of treatment was registered on an ordinal scale with four points: 1= No diagnosis of SAHS and patient is discharged; 2= Mild SAHS, patient should follow a conservative treatment and clinical control; 3= Moderate to severe SAHS, patient should begin continuous positive air pressure (CPAP) treatment; 4= Other sleep disorders are diagnosed (RC), or there is a need for full-night PSG owing to a discordance between clinical features and respiratory polygraphy in NRC. The indication for CPAP treatment followed the national-SEPAR guidelines summarized as: 1) Patients with severe SAHS-related symptoms with an AHI>10; or 2) Patients with mild to moderate clinical symptoms with an AHI>30. The human ethics committee of our hospital approved the protocol and informed consent was obtained from all the patients. Sleep studies: Reference hospital: Full-night polysomnography was performed in the usual manner. Briefly, the variables registered were electroencephalogram, chin electromyogram, electro-oculogram, tibial electromyogram, arterial oxygen saturation, ribcage and abdominal motion and their sum. Airflow was measured by cannula/thermistor. An apnea was defined as the absence or airflow equal to or greater than 10 seconds. Hypopnoea was defined by any discernible reduction in the amplitude of the airflow signal ending in an arousal and/or association with a 3% desaturation, with a duration of at least 10 seconds. An expert technician scored sleep stages and respiratory variables manually. An apnea-hypopnoea index (AHI) equal to or greater than 10 was considered abnormal.Non-reference centres: patients received a respiratory poligraphy with recording of body position, ribcage and abdominal motion, snoring, arterial oxygen saturation and airflow using a cannula/thermistor. The respiratory physician performed a manual scoring of the recording. The definitions of hypopnoea and apnea resembled those mentioned above, except in the case of arousal. Data analysis: Data were entered using SPSS 10.0 and imported to STATA 7.0 to perform the analysis (StatatCorp. 1999. Stata Statistical software: Release 7.0. College Station, TX: Stata Corporation). Descriptive analysis: Data were expressed as mean ± SD or percentage for quantitative and qualitative variables, respectively. For continuum variables, a logarithmic transformation was undertaken to normalise the distribution, if necessary. If the distribution was not symmetrical, data were expressed as percentiles. Concordance analysis: Evaluation of the concordance of the final outcome and the choice of treatment, between the RF and the NFC centres, was performed by using the statistic Kappa balanced, penalizing extreme discrepancies, following the classification of Landis & Koch (25). This procedure was also used for the concordance in the result of the AHI of the sleep study, categorised as follows: <10, 10-29, ≥30. Concordance in the results of the sleep study (AHI and CT90) was evaluated in accordance with the Band & Altman methodology and the concordance coefficient of Lin.

ELIGIBILITY:
Inclusion Criteria:

* Supected sleep apnea

Exclusion Criteria:

* Major diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2000-01; Study Completion 2004-04

PRIMARY OUTCOMES:
Concordance in sleep apnea management between reference vs non reference centres

SECONDARY OUTCOMES:
Concordane betwen polysomnographic data

CONTACTS AND LOCATIONS:
Overall Officials: Josep Montserrat, MD, Study Director — Fundacio Clinic. IDIBAPS
Locations (2):
- Spain (2):
  - Hospital Clinic. Fundacio Clinic.IDIBAPS, Barcelona
  - Hospital Clinic.Fundacio Clinic.IDIBAPS, Barcelona

REFERENCES:
- [Derived] Hernandez L, Torrella M, Roger N, Llunell A, Ballester E, Quinto L, Serrano M, Masa F, Montserrat JM. Management of sleep apnea: concordance between nonreference and reference centers. Chest. 2007 Dec;132(6):1853-7. doi: 10.1378/chest.07-0250. Epub 2007 Oct 9. PMID 17925431